CLINICAL TRIAL: NCT03905772
Title: Neuromuscular Adaptations After Training With Neuromuscular Electrical Stimulation Applied Over Nerve Trunk Compared With a Muscle Belly of Triceps Surae: Randomized Controlled Trial
Brief Title: Neuromuscular Adaptations After Training in the Muscle Belly of Triceps Surae
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Dr. Karenina has to change for another projetct due to Covid pandemic.
Sponsor: University of Brasilia (Other)
Collaborators: University of Burgundy (Other)
Responsible Party: Principal Investigator, João Luiz Q. Durigan, Physical Therapist Assistant Professor, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01326818.8.0000.8093
Record Dates: First submitted 2019-03-11; First posted 2019-04-05 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Electrical Stimulation
Keywords: Electrical stimulation; M wave; H reflex; Wide pulse

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Voluntary exercise (Experimental): The participants will perform 36 voluntary contractions of 20% of maximal voluntary isometrical contraction, 3 times per week for 8 weeks.
  Interventions: Other: Voluntary exercise
- Wide pulse responder group (Experimental): The participants will perform 36 contractions with the following current parameters: pulsed current (100 Hz, pulse duration 1 ms, Ton: 6 s, Toff: 18 s), 3 times per week for 8 weeks.
  This group will classified in responder in the acute fase.
  Interventions: Other: Wide pulse responder group
- Wide pulse non responder group (Experimental): The participants will perform 36 contractions with the following current parameters: pulsed current (100 Hz, pulse duration 1 ms, Ton: 6 s, Toff: 18 s), 3 times per week for 8 weeks.
  This group will classified in non responder in the acute fase.
  Interventions: Other: Wide pulse non responder group
- Pulsed current group (Experimental): The participants will perform 36 contractions with the following current parameters: pulsed current (100 Hz, pulse duration 250 μs, Ton: 6 s, Toff: 18 s), 3 times per week for 8 weeks.
  Interventions: Other: Pulsed current group

INTERVENTIONS:
Other: Voluntary exercise — The participants will perform 36 maximal voluntary contractions, 3 times per week for 8 weeks.
  Arms: Voluntary exercise
Other: Wide pulse responder group — The participants will perform 36 contractions with the following current parameters: pulsed current (100 Hz, pulse duration 1 ms, Ton: 6 s, Toff: 18 s), 3 times per week for 8 weeks. This group will be classified in responder group in acute fase.
  Arms: Wide pulse responder group
Other: Wide pulse non responder group — The participants will perform 36 contractions with the following current parameters: pulsed current (100 Hz, pulse duration 1 ms, Ton: 6 s, Toff: 18 s), 3 times per week for 8 weeks. This group will be classified in non responder group in acute fase.
  Arms: Wide pulse non responder group
Other: Pulsed current group — The participants will perform 36 contractions with the following current parameters: pulsed current (100 Hz, pulse duration 250 μs, Ton: 6 s, Toff: 18 s), 3 times per week for 8 weeks.
  Arms: Pulsed current group

SUMMARY:
This study aims to evaluate on an acute session of the central and peripheral contributions of electrical stimulation on the muscle belly of the triceps surae, electrical stimulation of the tibial nerve and voluntary exercise of the triceps surae muscle, and identify responders individuals and non-responders to stimulation of the tibial nerve. Another objective of the study is to compare the effects of conventional electrical stimulation applied to the sciatic triceps muscle, tibial nerve stimulation and voluntary exercise after eight weeks of training in healthy individuals.

DETAILED DESCRIPTION:
A controlled randomized controlled trial will be carried out by university students, divided equally into four groups: control group (GC), long responding pulse group (PLR), non-responder long pulse group (PLNR) and pulsed current group (CP) after the acute fase of the protocol. Muscular architecture (muscle thickness, pennation angle and fascicle length) of the muscles composing the sural triceps, H-reflex and M-wave tests (central and peripheral contribution), electromyographic signals of the medial and lateral gastrocnemius muscles and sole, voluntary and evoked joint torque of the muscles composing the sural triceps and level of sensorial discomfort. The independent intervention with the neuromuscular electrical stimulation and the isometric exercises performed by the control group will be considered as an independent variable. All groups will have the dependent variables evaluated 6 times, before, during and after the intervention, which will consist of 24 sessions (8 weeks). The training with neuromuscular electrical stimulation (NMES) will be performed 3 times a week and will never be applied for two consecutive days, as well as the voluntary exercises performed by the control group.

ELIGIBILITY:
Inclusion Criteria:

* Classified as physically active according to the INTERNATIONAL QUESTIONNAIRE OF PHYSICAL ACTIVITY,
* To practice only recreational physical activity,
* Achieve minimum torque of 30% of the (maximal voluntary isometric contraction during conventional NMES
* Be at least 3 months without practicing strength training.

Exclusion Criteria:

* Present some type of skeletal muscle dysfunction that may interfere with the tests,
* Present intolerance to NMES in the muscular or tibial nerve, Make use of analgesics, antidepressants, tranquillizers or other agents of central action
* To present cardiovascular or peripheral vascular problems, chronic diseases, neurological or muscular affections that will undermine the complete execution of the study design by the volunteer.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Central contribution (H reflex) after 15 minutes of acute session of electrical stimulation. | Baseline and after 15 minutes of electrical stimulation in the acute session.
  Central contribution will be measured before and after 15 minutes (36 contractions) of electrical stimulation in the acute session.
Change from Baseline Central contribution (H reflex) after 8 weeks of training with electrical stimulation. | Baseline and after 8 weeks of training with electrical stimulation.
  Central contribution will be measured before and after 8 weeks of training with electrical stimulation.
Change from Baseline Peripheral contribution (M wave) after 15 minutes of acute session of electrical stimulation | Baseline and after 15 minutes of electrical stimulation in the acute session
  Peripheral contribution will be measured before and after acute session 15 minutes (36 contractions) of electrical stimulation in the acute session.
Change from Baseline Peripheral contribution (M wave) after 8 weeks of traning with electrical atimulation | Baseline and after 8 weeks of training with electrical stimulation
  Peripheral contribution will be measured before and after 8 weeks of training with electrical stimulation.
Change from Baseline Voluntary torque after 8 weeks of training with electrical stimulation | Baseline and after 8 weeks of training with electrical stimulation
  Voluntary torque will be evaluated by an isokinetic dynamometer before and after an 8-week training period with electrical stimulation.
Change from Baseline Electromyographic signals after 8 weeks of training with electrical stimulation | Baseline and after 8 weeks of training with electrical stimulation
  Electromyographic signals will be evaluated by an electromyography before and after an 8-week training period with electrical stimulation.

SECONDARY OUTCOMES:
Change from Baseline Evoked torque after 8 weeks of training with electrical stimulation | Baseline and after 8 weeks of training with electrical stimulation
  Evoked torque will be evaluated by an isokinetic dynamometer before and after an 8-week training period with electrical stimulation.
Change from Baseline Discomfort sensory after 8 weeks of training with electrical stimulation | Baseline and after 8 weeks of training with electrical stimulation
  Discomfort sensory will be evaluated by Visual Analogic Scale before and after an 8-week training period with electrical stimulation. The Visual Analogic Scale assess pain by rating the subjective perceived disconfort of the subject from 0 (no pain) to 10 (unbearable pain)

CONTACTS AND LOCATIONS:
Overall Officials: João Durigan, PhD, Study Director — University of Brasilia
Locations (1):
- Faculty of Ceilandia UnB, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dirks ML, Hansen D, Van Assche A, Dendale P, Van Loon LJ. Neuromuscular electrical stimulation prevents muscle wasting in critically ill comatose patients. Clin Sci (Lond). 2015 Mar;128(6):357-65. doi: 10.1042/CS20140447. PMID 25296344
- [Result] Chae J, Sheffler L, Knutson J. Neuromuscular electrical stimulation for motor restoration in hemiplegia. Top Stroke Rehabil. 2008 Sep-Oct;15(5):412-26. doi: 10.1310/tsr1505-412. PMID 19008202
- [Result] Brocherie F, Babault N, Cometti G, Maffiuletti N, Chatard JC. Electrostimulation training effects on the physical performance of ice hockey players. Med Sci Sports Exerc. 2005 Mar;37(3):455-60. doi: 10.1249/01.mss.0000155396.51293.9f. PMID 15741845
- [Result] Billot M, Martin A, Paizis C, Cometti C, Babault N. Effects of an electrostimulation training program on strength, jumping, and kicking capacities in soccer players. J Strength Cond Res. 2010 May;24(5):1407-13. doi: 10.1519/JSC.0b013e3181d43790. PMID 20386476
- [Result] Medeiros FV, Bottaro M, Vieira A, Lucas TP, Modesto KA, Bo APL, Cipriano G Jr, Babault N, Durigan JLQ. Kilohertz and Low-Frequency Electrical Stimulation With the Same Pulse Duration Have Similar Efficiency for Inducing Isometric Knee Extension Torque and Discomfort. Am J Phys Med Rehabil. 2017 Jun;96(6):388-394. doi: 10.1097/PHM.0000000000000631. PMID 27680427
- [Result] Vaz MA, Baroni BM, Geremia JM, Lanferdini FJ, Mayer A, Arampatzis A, Herzog W. Neuromuscular electrical stimulation (NMES) reduces structural and functional losses of quadriceps muscle and improves health status in patients with knee osteoarthritis. J Orthop Res. 2013 Apr;31(4):511-6. doi: 10.1002/jor.22264. Epub 2012 Nov 8. PMID 23138532
- [Result] Gondin J, Brocca L, Bellinzona E, D'Antona G, Maffiuletti NA, Miotti D, Pellegrino MA, Bottinelli R. Neuromuscular electrical stimulation training induces atypical adaptations of the human skeletal muscle phenotype: a functional and proteomic analysis. J Appl Physiol (1985). 2011 Feb;110(2):433-50. doi: 10.1152/japplphysiol.00914.2010. Epub 2010 Dec 2. PMID 21127206
- [Result] Ward AR, Robertson VJ. The variation in fatigue rate with frequency using kHz frequency alternating current. Med Eng Phys. 2000 Nov;22(9):637-46. doi: 10.1016/s1350-4533(00)00085-0. PMID 11259932
- [Result] Ward AR, Chuen WL. Lowering of sensory, motor, and pain-tolerance thresholds with burst duration using kilohertz-frequency alternating current electric stimulation: part II. Arch Phys Med Rehabil. 2009 Sep;90(9):1619-27. doi: 10.1016/j.apmr.2009.02.022. PMID 19735792
- [Result] Ward AR, Robertson VJ, Ioannou H. The effect of duty cycle and frequency on muscle torque production using kilohertz frequency range alternating current. Med Eng Phys. 2004 Sep;26(7):569-79. doi: 10.1016/j.medengphy.2004.04.007. PMID 15271284
- [Result] Paillard T, Noe F, Bernard N, Dupui P, Hazard C. Effects of two types of neuromuscular electrical stimulation training on vertical jump performance. J Strength Cond Res. 2008 Jul;22(4):1273-8. doi: 10.1519/JSC.0b013e3181739e9c. PMID 18545178
- [Result] Filipovic A, Kleinoder H, Dormann U, Mester J. Electromyostimulation--a systematic review of the influence of training regimens and stimulation parameters on effectiveness in electromyostimulation training of selected strength parameters. J Strength Cond Res. 2011 Nov;25(11):3218-38. doi: 10.1519/JSC.0b013e318212e3ce. PMID 21993042
- [Result] Filipovic A, Kleinoder H, Dormann U, Mester J. Electromyostimulation--a systematic review of the effects of different electromyostimulation methods on selected strength parameters in trained and elite athletes. J Strength Cond Res. 2012 Sep;26(9):2600-14. doi: 10.1519/JSC.0b013e31823f2cd1. PMID 22067247
- [Result] Selkowitz DM, Rossman EG, Fitzpatrick S. Effect of burst-modulated alternating current carrier frequency on current amplitude required to produce maximally tolerated electrically stimulated quadriceps femoris knee extension torque. Am J Phys Med Rehabil. 2009 Dec;88(12):973-8. doi: 10.1097/PHM.0b013e3181c1eda5. PMID 19935181
- [Result] Binder-Macleod SA, Halden EE, Jungles KA. Effects of stimulation intensity on the physiological responses of human motor units. Med Sci Sports Exerc. 1995 Apr;27(4):556-65. PMID 7791587
- [Result] Gorgey AS, Black CD, Elder CP, Dudley GA. Effects of electrical stimulation parameters on fatigue in skeletal muscle. J Orthop Sports Phys Ther. 2009 Sep;39(9):684-92. doi: 10.2519/jospt.2009.3045. PMID 19721215
- [Result] Gorgey AS, Dudley GA. The role of pulse duration and stimulation duration in maximizing the normalized torque during neuromuscular electrical stimulation. J Orthop Sports Phys Ther. 2008 Aug;38(8):508-16. doi: 10.2519/jospt.2008.2734. Epub 2008 Aug 1. PMID 18678958
- [Result] Bax L, Staes F, Verhagen A. Does neuromuscular electrical stimulation strengthen the quadriceps femoris? A systematic review of randomised controlled trials. Sports Med. 2005;35(3):191-212. doi: 10.2165/00007256-200535030-00002. PMID 15730336
- [Result] Ward AR, Oliver WG, Buccella D. Wrist extensor torque production and discomfort associated with low-frequency and burst-modulated kilohertz-frequency currents. Phys Ther. 2006 Oct;86(10):1360-7. doi: 10.2522/ptj.20050300. PMID 17012640
- [Result] Laufer Y, Elboim M. Effect of burst frequency and duration of kilohertz-frequency alternating currents and of low-frequency pulsed currents on strength of contraction, muscle fatigue, and perceived discomfort. Phys Ther. 2008 Oct;88(10):1167-76. doi: 10.2522/ptj.20080001. Epub 2008 Aug 14. PMID 18703676
- [Result] Dantas LO, Vieira A, Siqueira AL Jr, Salvini TF, Durigan JL. Comparison between the effects of 4 different electrical stimulation current waveforms on isometric knee extension torque and perceived discomfort in healthy women. Muscle Nerve. 2015 Jan;51(1):76-82. doi: 10.1002/mus.24280. PMID 24809656
- [Result] Bergquist AJ, Wiest MJ, Collins DF. Motor unit recruitment when neuromuscular electrical stimulation is applied over a nerve trunk compared with a muscle belly: quadriceps femoris. J Appl Physiol (1985). 2012 Jul;113(1):78-89. doi: 10.1152/japplphysiol.00074.2011. Epub 2012 May 3. PMID 22556395
- [Result] Maffiuletti NA. Physiological and methodological considerations for the use of neuromuscular electrical stimulation. Eur J Appl Physiol. 2010 Sep;110(2):223-34. doi: 10.1007/s00421-010-1502-y. Epub 2010 May 15. PMID 20473619
- [Result] Barss TS, Ainsley EN, Claveria-Gonzalez FC, Luu MJ, Miller DJ, Wiest MJ, Collins DF. Utilizing Physiological Principles of Motor Unit Recruitment to Reduce Fatigability of Electrically-Evoked Contractions: A Narrative Review. Arch Phys Med Rehabil. 2018 Apr;99(4):779-791. doi: 10.1016/j.apmr.2017.08.478. Epub 2017 Sep 19. PMID 28935232
- [Result] Gregory CM, Bickel CS. Recruitment patterns in human skeletal muscle during electrical stimulation. Phys Ther. 2005 Apr;85(4):358-64. PMID 15794706
- [Result] Bergquist AJ, Clair JM, Collins DF. Motor unit recruitment when neuromuscular electrical stimulation is applied over a nerve trunk compared with a muscle belly: triceps surae. J Appl Physiol (1985). 2011 Mar;110(3):627-37. doi: 10.1152/japplphysiol.01103.2010. Epub 2010 Dec 23. PMID 21183628
- [Result] Bergquist AJ, Clair JM, Lagerquist O, Mang CS, Okuma Y, Collins DF. Neuromuscular electrical stimulation: implications of the electrically evoked sensory volley. Eur J Appl Physiol. 2011 Oct;111(10):2409-26. doi: 10.1007/s00421-011-2087-9. Epub 2011 Jul 30. PMID 21805156
- [Result] da Silva VZ, Durigan JL, Arena R, de Noronha M, Gurney B, Cipriano G Jr. Current evidence demonstrates similar effects of kilohertz-frequency and low-frequency current on quadriceps evoked torque and discomfort in healthy individuals: a systematic review with meta-analysis. Physiother Theory Pract. 2015;31(8):533-9. doi: 10.3109/09593985.2015.1064191. Epub 2015 Oct 14. PMID 26467544
- [Result] Maffiuletti NA, Cometti G, Amiridis IG, Martin A, Pousson M, Chatard JC. The effects of electromyostimulation training and basketball practice on muscle strength and jumping ability. Int J Sports Med. 2000 Aug;21(6):437-43. doi: 10.1055/s-2000-3837. PMID 10961520
- [Result] Flann KL, LaStayo PC, McClain DA, Hazel M, Lindstedt SL. Muscle damage and muscle remodeling: no pain, no gain? J Exp Biol. 2011 Feb 15;214(Pt 4):674-9. doi: 10.1242/jeb.050112. PMID 21270317
- [Result] Jenkins NDM, Miramonti AA, Hill EC, Smith CM, Cochrane-Snyman KC, Housh TJ, Cramer JT. Greater Neural Adaptations following High- vs. Low-Load Resistance Training. Front Physiol. 2017 May 29;8:331. doi: 10.3389/fphys.2017.00331. eCollection 2017. PMID 28611677
- [Result] Oliveira P, Modesto KAG, Bottaro M, Babault N, Durigan JLQ. Training Effects of Alternated and Pulsed Currents on the Quadriceps Muscles of Athletes. Int J Sports Med. 2018 Jul;39(7):535-540. doi: 10.1055/a-0601-6742. Epub 2018 May 22. PMID 29788511
- [Result] Blazevich AJ, Gill ND, Zhou S. Intra- and intermuscular variation in human quadriceps femoris architecture assessed in vivo. J Anat. 2006 Sep;209(3):289-310. doi: 10.1111/j.1469-7580.2006.00619.x. PMID 16928199
- [Result] Morse CI, Thom JM, Birch KM, Narici MV. Changes in triceps surae muscle architecture with sarcopenia. Acta Physiol Scand. 2005 Mar;183(3):291-8. doi: 10.1111/j.1365-201X.2004.01404.x. PMID 15743389
- [Result] Grospretre S, Jacquet T, Lebon F, Papaxanthis C, Martin A. Neural mechanisms of strength increase after one-week motor imagery training. Eur J Sport Sci. 2018 Mar;18(2):209-218. doi: 10.1080/17461391.2017.1415377. Epub 2017 Dec 17. PMID 29249176
- [Result] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Result] Duclay J, Martin A. Evoked H-reflex and V-wave responses during maximal isometric, concentric, and eccentric muscle contraction. J Neurophysiol. 2005 Nov;94(5):3555-62. doi: 10.1152/jn.00348.2005. Epub 2005 Jul 27. PMID 16049144
- [Result] Babault N, Pousson M, Michaut A, Van Hoecke J. Effect of quadriceps femoris muscle length on neural activation during isometric and concentric contractions. J Appl Physiol (1985). 2003 Mar;94(3):983-90. doi: 10.1152/japplphysiol.00717.2002. Epub 2002 Nov 15. PMID 12571130
- [Result] Kent-Braun JA. Central and peripheral contributions to muscle fatigue in humans during sustained maximal effort. Eur J Appl Physiol Occup Physiol. 1999 Jun;80(1):57-63. doi: 10.1007/s004210050558. PMID 10367724
- [Result] Pajoutan M, Ghesmaty Sangachin M, Cavuoto LA. Central and peripheral fatigue development in the shoulder muscle with obesity during an isometric endurance task. BMC Musculoskelet Disord. 2017 Jul 21;18(1):314. doi: 10.1186/s12891-017-1676-0. PMID 28732481
- [Result] Botter A, Oprandi G, Lanfranco F, Allasia S, Maffiuletti NA, Minetto MA. Atlas of the muscle motor points for the lower limb: implications for electrical stimulation procedures and electrode positioning. Eur J Appl Physiol. 2011 Oct;111(10):2461-71. doi: 10.1007/s00421-011-2093-y. Epub 2011 Jul 28. PMID 21796408